CLINICAL TRIAL: NCT01613144
Title: Expandable Pedicle Screws Versus Fenestrated Pedicle Screws Augmented With Polymethylmethacrylate (PMMA): Complications and Clinical Outcomes in Patients With Osteoporosis or Poor Bone Quality
Brief Title: OsseoScrew Versus Fenestrated Pedicle Screws Augmented With Polymethylmethacrylate
Acronym: EVOLVE
Status: Completed | Type: Observational
Sponsor: Alphatec Spine, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: REC-000784
Record Dates: First submitted 2012-05-31; First posted 2012-06-07 (Estimated); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Osteoporosis; Poor Bone Quality
Keywords: Osteopenia; Stenosis; Instability; Tumor
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Constriction, Pathologic; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- OsseoScrew: Test Product: OsseoScrew Spinal Fixation System
  Interventions: Device: OsseoScrew Spinal Fixation System
- Fenestrated Screw: Control Product: Any commercially available fenestrated screw system augmented with PMMA

INTERVENTIONS:
Device: OsseoScrew Spinal Fixation System — Surgical intervention
  Groups: OsseoScrew

SUMMARY:
The purpose of this clinical investigation was to collect clinical evidence of the safety and efficacy of the OsseoScrew System. The OsseoScrew System is intended to provide immobilization and stabilization of spinal segments in skeletally mature patients as an adjunct to fusion. The study was designed to compare the safety and efficacy of OsseoScrew compared to any other commercially available fenestrated pedicle screw system augmented with PMMA for posterior spinal fixation after surgical correction of spinal deformity or pathology.

DETAILED DESCRIPTION:
This was a randomized, open-label, controlled, multi-center study in which patients were randomized in a 1:1 ratio to receive either the OsseoScrew or any commercially available fenestrated screw augmented with polymethylmethacrylate (PMMA) (Control group) for posterior spinal fixation after surgical correction of spinal deformity or pathology. The study was planned to include up to 150 skeletally mature patients with spinal instability and osteopenia at up to 10 sites. Patients were to return postoperatively at 6 weeks (± 2 weeks) and at 6, 12, and 24 months (± 2 months) for assessments.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Spinal instability or deformity requiring fusion with instrumentation
3. Osteopenia defined as (T-Score of less than -1.0)
4. No response to nonoperative treatment modalities preceding enrollment.
5. Subject is willing and able to provide informed consent and agrees to release medical information for purposes of this study and to return for scheduled follow-up evaluations

Exclusion Criteria:

1. Active systemic or local infection
2. A life expectancy less than the study duration
3. Autoimmune disorders
4. Currently an alcohol, solvent, or drug abuser
5. Psychiatric or cognitive impairment that, in the opinion of the investigator, would interfere with the subject's ability to comply with the study requirements
6. History of allergies to any of the device components including but not limited to commercially pure titanium, titanium alloy, polymethylmethacrylate or Zirconium Oxide (ZrO2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 skeletally mature study subjects with spinal instability and osteopenia will be enrolled in the study. Subjects will be randomized 1:1 to the OsseoScrew or the control group.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2012-05; Primary Completion 2017-02-12 (Actual); Study Completion 2017-11-08 (Actual)

PRIMARY OUTCOMES:
Safety Endpoint: Rate of device-related or PMMA-related complications | 24 months
  The proportion of patients who were free from device-related or PMMA-related complications leading to revision, supplemental fixation, non-elective removal, or reoperation throughout the study. Complications included, but were not limited to device or PMMA fracture, device or PMMA-related loosening, device or PMMA-related device disassembly, device migration or PMMA extravasation.
Efficacy Endpoint: Successful radiographic fusion | 24 months
  Presence of continuous bridging bone across the implant

SECONDARY OUTCOMES:
Oswestry Disability Index | 24 months
  This is a measure of the patient's self reported permanent functional disability. Each section is scored on a 1-5 scale with 5 representing the greatest disability.
Visual Analogue Scale for back pain | 24 months
  This is a measure of the characteristic or attitude that is believed to range across a continuum of values to measure pain intensity. The range of score is from 0 - 100. The patient marks on the line the point that they feel represents their perception of their current state. A higher score indicates greater pain intensity.
Adverse events | 24 months
  Adverse event rates

CONTACTS AND LOCATIONS:
Overall Officials: Bita Ghadimi, Study Director — Alphatec Spine, Inc.
Locations (10):
- Belgium (4):
  - O.L. Vrouwziekenhuis, Aalst
  - CHIREC du Clinique, Brussels
  - ULB Hopital Erasme, Brussels
  - CHC St. Joseph, Liège
- Germany (2):
  - Katholisches Klinikum Koblenz - Montabaur/, Koblenz
  - University Medical Center Mainz/, Mainz
- San Giovanni Addolorata Hospital, Rome, Italy
- Spain (2):
  - Institut d'Assistència Sanitària, Girona
  - Hospital de Leon, León
- The Royal National Orthopaedic Hospital, Stanmore, United Kingdom

IPD SHARING:
Plan to Share IPD: No